CLINICAL TRIAL: NCT02222194
Title: Assessment of Surgical Mediastinal sTaging in cN1 Lung canceR
Brief Title: The Value of Surgical Mediastinal Staging in Clinical N1 Lung Cancer
Acronym: ASTER3
Status: Completed | Type: Observational
Sponsor: Johnny Moons (Other)
Responsible Party: Sponsor-Investigator, Johnny Moons, Data Manager / Clinical Trial Coordinator, University Hospital, Gasthuisberg
Organization: University Hospital, Gasthuisberg (Other)
Other Study IDs: ASTER 3
Record Dates: First submitted 2014-08-18; First posted 2014-08-21 (Estimated); Last update posted 2017-07-25 (Actual); Status verified 2017-07

CONDITIONS: Non Small Cell Lung Cancer
Keywords: Lung cancer; Surgery; Videomediastinoscopy
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Lung Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- VAM: Patients with operable and resectable cT1-2-selected T3 cN1cM0 NSCLC undergo VAM for mediastinal lymph node staging. After VAM, patients without tissue proof of N2/3 disease at surgical staging undergo a VATS or thoracotomy with systematic lymph node dissection during the same anaesthesia or at a later stage.
  Sensitivity, NPV and accuracy of staging with VAM will be calculated. Provided N2 lymph node metastases are proven by VAM the patient goes off study protocol and can further be assessed/treated according to local clinical practice.

SUMMARY:
In case of PET or CT based cN1 (suspected) NSCLC, ESTS guidelines propose mediastinal staging by echo-endoscopy OR mediastinoscopy. Recent data show a sensitivity of less than 50% for echo-endoscopy to detect N2 disease in cN1 NSCLC patients, while prevalence of mediastinal nodal disease was 24% (unpublished data Aster II).2 The investigators plan to perform a prospective multicentric observational study to measure the sensitivity of mediastinal staging by video-assisted mediastinoscopy (VAM) in cN1 operable and resectable (suspected) NSCLC patients.

DETAILED DESCRIPTION:
Few reports in the literature evaluated the final pathological stage distribution of patients with resectable and operable non-small cell lung cancer (NSCLC) with clinical stage cN1. These retrospective series demonstrated that patients with computed tomography (CT) based cN1 often had clinically occult mediastinal lymph node metastases (N2/3 disease). Hishida et al. reported that 30% of 143 patients with cN1 were diagnosed N2/3 by mediastinoscopy3. Watanabe et al. reported that 37% of 168 patients with cN1 were diagnosed N2/3 by mediastinoscopy 4. Adding FDG-positron emission tomography (PET) to CT might enable the detection of N2/3 disease among these cN1 patients, but negative PET findings do not necessarily exclude N2/3 disease. Kim et al reported that 19,2 % of 99 patients with cN1, in whom cN2 was ruled out by PET-CT scan, were found to have pathologic N2 disease at pulmonary resection with mediastinal lymph node dissection.5 In conclusion, 20-30% of patients with cN1 nodes on imaging, and normal sized FDG-negative mediastinal lymph nodes on CT and PET have malignant involvement in their mediastinal nodes.

The ACCP guidelines state that invasive preoperative mediastinal staging should be performed in these cN1 patients 6. The updated ESTS guidelines recommend mediastinal staging by echo-endoscopic or mediastinoscopy.1 Non-randomized trials suggested the potential of linear endosonography for mediastinal staging 7-9. However, the patients with cN1 disease form only a minority in these studies. A recently performed prospective ASTER 2 trial (N=100) showed a sensitivity of echo-endoscopic for mediastinal staging of 38% (ITT analysis), while the prevalence of mediastinal nodal disease was 24% (unpublished data Aster 2) 2. The conclusion made by ASTER 2 is that a negative endosonography must be followed by a VAM. However, the investigators consider such double approach not cost-effective in a setting with N2 prevalence <30%. Therefore, it seems reasonable to perform a VAM instead of an endosonography in cN1 patients, which is one of the proposed strategies in the recent ESTS guidelines.1 However, there is no prospective study to date that assessed the sensitivity, NPV and accuracy of VAM in a well-defined group of cN1 patients.

Several publications have demonstrated a lobe-specific mediastinal nodal drainage for upper versus lower lobe NSCLC. Shapiro et al conclude that in early lung cancer, including cN1 disease, lobe-specific mediastinal dissection is warranted 10. However, in this study the only patient with a positive subcarinal node, upper lobe tumour, and negative superior mediastinal nodes had positive N1 nodes. To the investigators knowledge there is no study focussing on mediastinal nodal dissemination patterns in cN1 patients.

ELIGIBILITY:
Inclusion Criteria:

(Suspected) NSCLC Medical operable and surgical resectable cT1, cT2 selected cT3 (i.e. intraparenchymal tumour >7cm, T3 chest wall, or T3 based on additional nodule in the lobe of the primary tumour) cN1 based on CT or PET 18 years or older Informed Consent

Exclusion Criteria:

History of mediastinoscopy No integrated FDG PET/CT available No videomediastinoscopy available EBUS/EUS for mediastinal staging of present N1 disease cN2: mediastinal nodes enlarged on CT or Pet positive invasion of mediastinal pleura invasion of phrenic nerve invasion of parietal pericardium tumour in main bronchus less than 2cm form the main carina cT4 cM1 former therapy for lung cancer (chemotherapy, radiotherapy, surgery) technical contraindication for videomediastinoscopy ( eg extreme kyphosis, cutaneous tracheostomy, extreme goiter) pregnancy inability to consent

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with operable and resectable cT1-2- selectedT3 cN1 (suspected) NSCLC. (selected T3 = intraparenchymal tumour >7cm or T3 chest wall or T3 additional nodule, excluding mediastinal invasion or invasion of the main bronchus < 2cm from the carina)
Sampling Method: Probability Sample
Enrollment: 105 (Actual)
Dates: Start 2014-08; Primary Completion 2017-03 (Actual); Study Completion 2017-05-30 (Actual)

PRIMARY OUTCOMES:
Sensitivity of VAM | at surgery (VAM)
  Sensitivity (%) of surgical mediastinal staging by video-assisted mediastinoscopy in clinical N1; true positives (TP) = cN1 and pN1 - false negatives (FP) = cN1 and pN2/3; sensitivity is calculated as TP / (TP+FN)

SECONDARY OUTCOMES:
Prevalence of N2/3 disease after VAM | at surgery (VAM)
  % of patients with cN1 disease who show pN2/3 disease after VAM

CONTACTS AND LOCATIONS:
Overall Officials: Herbert Decaluwé, MD, Study Director — Universitaire Ziekenhuizen KU Leuven
Locations (10):
- University Hospital Leuven, Leuven, Belgium
- Aix-Marseille University & Hospitals System of Marseille (AP-HM), Marseille, France
- Germany (4):
  - ELK Berlin Chest Hospital, Berlin
  - Albert-Ludwigs-University Freiburg, Freiburg im Breisgau
  - Katholisches Klinikum Koblenz, Koblenz
  - Katholisches Klinikum, Thoraxchirurgie, Koblenz
- Spain (2):
  - Hospital Universitari Mutua Terrassa, Barcelona
  - Hospital Clinic; Barcelona University, Barcelona
- University Hospital, Division of Thoracic Surgery, Zurich, Switzerland
- Istanbul University, Cerrahpasa Medical Faculty, Istanbul, Turkey (Türkiye)

REFERENCES:
- [Derived] Decaluwe H, Dooms C, D'Journo XB, Call S, Sanchez D, Haager B, Beelen R, Kara V, Klikovits T, Aigner C, Tournoy K, Zahin M, Moons J, Brioude G, Trujillo JC, Klepetko W, Turna A, Passlick B, Molins L, Rami-Porta R, Thomas P, Leyn P. Mediastinal staging by videomediastinoscopy in clinical N1 non-small cell lung cancer: a prospective multicentre study. Eur Respir J. 2017 Dec 21;50(6):1701493. doi: 10.1183/13993003.01493-2017. Print 2017 Dec. PMID 29269579